CLINICAL TRIAL: NCT04066114
Title: Regulatory T Cell Modulation in Kidney Transplantation With Biologic Blockade of Dual Effector Pathways, CD28 and IL-6 (CTOT-24)
Brief Title: Treg Modulation With CD28 and IL-6 Receptor Antagonists
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOT-24; NIAID CRMS ID#: 38581 (Other: DAIT NIAID)
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Living-Donor Kidney Transplant; Kidney Transplant Recipients
Keywords: adult living-donor kidney transplant recipients; novel immunosuppressive (IS) therapy regimen; lulizumab pegol (BMS-931699); CD28 and IL-6 biologic blockade; CD28 and IL-6 receptor antagonists; T regulatory cells (Treg) modulation
MeSH Terms: interventions — lulizumab pegol; thymoglobulin; Methylprednisolone; Methylprednisolone Hemisuccinate; tocilizumab; Prednisone; Everolimus; Abatacept; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- lulizumab pegol + novel ISR (Experimental): lulizumab pegol + novel ISR: lulizumab pegol plus immunosuppressive regimen (anti-thymocyte globulin (rabbit), steroids,) belatacept, tocilizumab, and everolimus)
  Interventions: Biological: lulizumab pegol; Biological: antithymocyte globulin (rabbit); Drug: methylprednisolone; Biological: tocilizumab; Drug: Prednisone; Drug: everolimus; Biological: belatacept; Drug: mycophenolate mofetil; Drug: mycophenolic acid

INTERVENTIONS:
Biological: lulizumab pegol — 25 mg subcutaneously (SC) on Day 1 post transplantation then 12.5 mg SC weekly through day 77 (Week 11)
  Other Names: BMS-931699
Biological: antithymocyte globulin (rabbit) — Study participants are administered four doses of rabbit anti-thymocyte globulin, total dose 6 mg/kg given in divided doses on the day of transplantation and days 1-3.
  Other Names: ATG (rabbit); Thymoglobulin®
Drug: methylprednisolone — 500 mg (IV) on Day 0 (day of transplantation), 250 mg (IV) on Day 1 and 125 mg (IV) on Day 2
  Other Names: Solu-Medrol ®
Biological: tocilizumab — 8 mg/kg (IV) on Day 2 post transplantation followed by 162 mg (SC) every 2 weeks through day 168 (Week 24)
  Other Names: Actemra®
Drug: Prednisone — Beginning on Day 3 post transplantation, taken orally: 60 mg daily
  * Days 4 through 10: 30 mg daily
  * Days 11 through 17: 20 mg daily
  * Days 18 through 24: 10 mg daily
  * After Day 24: continued taper of dose to final maintenance dose of 5 mg, per protocol
  Other Names: prednisone tablets; Rayos®
Drug: everolimus — Initial dose of 0.75 mg taken orally twice daily on Day 14 days after transplantation. Dose will be titrated to target trough levels 3-8 ng/mL.
  Other Names: Zortress®
Biological: belatacept — 5 mg/kg (IV) every 4 weeks starting on Day 84 (Week 12) and continuing through Day 364 (Week 52)
  Other Names: Nulojix®
Drug: mycophenolate mofetil — mycophenolate mofetil is started no later than one day after transplant at 1000mg PO twice daily provided WBC count permits, staying on it until everoliumus level is within therapeutic range. Participants that do no tolerate everolimus can stay on or switch back to mycophenolate mofetil 1000 mg twice daily and remain in trial.
  Other Names: MMF; CellCept®
Drug: mycophenolic acid — mycophenolic acid is started no later than one day after transplant at 720mg PO twice daily provided WBC count permits, staying on it until everoliumus level is within therapeutic range. Participants that do not tolerate everolimus can stay on or switch back to 720 mg twice daily of mycophenolic acid and remain in trial.
  Other Names: Myfortic®

SUMMARY:
The purpose of this study is to evaluate the safety of using lulizumab pegol with tocilizumab, belatacept, and everolimus in kidney transplant recipients.

DETAILED DESCRIPTION:
This research study is for adults who are planning to have a kidney transplant from a living donor.

In Brief:

Those who have a transplant take immunosuppressive therapy to prevent the body from rejecting the transplanted organ. Rejection occurs when the body's defense system (immune cells) recognizes the transplant as a foreign object. These immune cells and the substances they produce can damage the transplanted kidney. It is important to prevent rejection episodes, so the kidney transplant lasts as long as possible.

Most transplant doctors in the United States give a combination of two or three drugs to prevent rejection. People with a transplant must take these drugs every day. Although kidney transplant recipients usually do well in the first five years after transplant, researchers want to find new ways to prevent rejection and avoid the side effects that the current drugs can cause.

This study will test a new combination of four drugs to evaluate whether this combination is safe for kidney transplant recipients:

* lulizumab pegol (BMS-931699)
* tocilizumab
* belatacept and
* everolimus.

Belatacept and everolimus are already approved for use as anti-rejection drugs in kidney transplant recipients. Lulizumab pegol and tocilizumab act on specific molecules (specifically CD28 and interleukin 6, respectively) on immune cells: these actions are different from how the older rejection drugs work.

Summary: This is a prospective multicenter open-label clinical trial of 10 living donor kidney transplant recipients. Safety of lulizumab pegol (BMS-931699) in the context of a novel immunosuppressive regimen (anti-thymocyte globulin (rabbit) (ATG), steroids,) Nulojix® (belatacept), Actemra® (tocilizumab), and Zortress®(everolimus)) will be assessed. Study participation involves a minimum of one year of follow-up post-transplant.

*** IMPORTANT NOTICE: *** The National Institute of Allergy and Infectious Diseases and the Clinical Trials in Organ Transplantation (CTOT) do not recommend the discontinuation of immunosuppressive therapy for recipients of cell, organ, or tissue transplants outside of physician-directed, controlled clinical studies. Discontinuation of prescribed immunosuppressive therapy can result in serious health consequences and should only be performed in certain rare circumstances, upon the recommendation and with the guidance of your health care provider.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all the following criteria are eligible for enrollment as study participants:

1. Able to understand and provide informed consent
2. Agreement to use highly effective (<1% failure rate) methods of contraception: Women of Childbearing Potential (WOCBP)-

   * Progestogen only hormonal contraception associated with inhibition of ovulation,
   * Hormonal methods of contraception including oral contraceptive pills containing a combination of estrogen + progesterone, vagina ring, injectables, implants and intrauterine devices (IUDs),
   * Non-hormonal IUDs,
   * Bilateral tubal occlusion,
   * Vasectomized partner,
   * Intrauterine hormone-releasing system (IUS), or
   * Complete abstinence.

   Note: Female participants of childbearing potential must consult with their physician and determine the most suitable method(s) from this list to be used for 12 months while on study drug regimen.

   Male Participants-

   --Must use a latex or other synthetic condom during any sexual activity with WOCBP until one month after the last dose of lulizumab (e.g., up to 3.5 months in duration).
3. Recipient of primary, nonhuman leukocyte antigen identical living donor kidney transplant
4. No donor specific antibodies prior to transplant that are considered to be of clinical significance by the site investigator
5. Epstein-Barr virus (EBV) positive serology
6. Cytomegalovirus (CMV) positive serology, unless donor-recipient pair are both CMV negative
7. Negative testing for latent Tuberculosis (TB) infection within 3 months prior to transplant

   * Testing should be conducted using either a purified protein derivative (PPD) or an interferon-gamma release assay blood test for TB (i.e. QuantiFERON®-TB Gold in-Tube test or T-SPOT® TB test)
   * Subjects with a positive test for latent TB infection must complete appropriate therapy for Latent tuberculosis infection (LTBI). ---A subject is considered eligible only if they have a negative test for LTBI within 3 months prior to transplant or, they have appropriately completed LTBI therapy prior to transplant.

   Note: Latent TB infection treatment regimens should be among those endorsed by the CDC (Division of TB Elimination, 2016).
8. In the absence of contraindication, vaccinations must be up to date for hepatitis B, influenza, pneumococcal, varicella and herpes zoster, and measles, mumps, and rubella (MMR)
9. Hepatitis C Virus (HCV) antibody positive subjects with negative HCV by PCR testing are eligible if they:

   * have spontaneously cleared infection, or
   * are in sustained virologic remission for at least 12 weeks after treatment for HCV.
10. Negative SARS-CoV-2 PCR test result performed within 2 weeks of transplant (SARS-CoV-2 is the virus that causes COVID-19)

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants-

1. Prisoners or subjects who are compulsorily detained
2. Inability or unwillingness of a participant to give written informed consent or comply with study protocol
3. Candidate for a multiple solid organ or tissue transplants
4. Prior history of organ or cellular transplantation
5. Known to have idiopathic focal segmental glomerulosclerosis (FSGS) as the underlying cause of kidney failure (ESRD)
6. Requirement for uninterrupted anticoagulation therapy, including Plavix.
7. Known hypersensitivity to mechanistic target of rapamycin (mTOR) inhibitors or contraindication to everolimus (including history of wound healing complications)
8. History of severe allergic and/or anaphylactic reactions to humanized or murine monoclonal antibodies
9. Hypersensitivity to rabbit proteins or rabbit anti-thymocyte Globulin (ATG)
10. Known hypersensitivity to ACTEMRA® (tocilizumab) or lulizumab pegol (BMS-931699)
11. The human immunodeficiency virus (HIV) infected subjects, including those who are well controlled on antiretrovirals
12. Positive hepatitis B surface antigen (HBSAg), or hepatitis B core antibody (HBcAB) serology
13. Hepatitis C virus antibody positive (HCV Ab+) subjects who have failed to demonstrate sustained viral remission for more than 12 weeks after anti-viral treatment
14. Subjects with a previous history of active Tuberculosis (TB)
15. Known active current viral, fungal, mycobacterial or other infections (including, but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster)
16. Donor or recipient residing in areas where the annual incidence ≥ 21 cases per 100,000) for coccidioidomycosis according to current CDC map: (https://www.cdc.gov/fungal/diseases/coccidioidomycosis/causes.html)

    * Donors or recipients residing in low risk zones (annual <21 cases per 100,000) will not require additional screening
17. History of malignancy except treated basal cell cancer of the skin
18. History of hemolytic-uremic syndrome/ thrombotic thrombocytopenia purpura
19. History of demyelinating disorders (e.g., multiple sclerosis, chronic inflammation demyelinating polyneuropathy)
20. History of gastrointestinal perforations, active inflammatory bowel disease or diverticulitis
21. Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation
22. Receipt of a live vaccine within 30 days prior to transplantation.
23. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may:

    * pose additional risks from participation in the study,
    * may interfere with the participant's ability to comply with study requirements, or
    * that may impact the quality or interpretation of the data obtained from the study
24. Severe hyperlipidemia (defined by total cholesterol >350 mg/dL, LDL >190 mg/dL, or triglycerides >500 mg/dL)
25. Transaminase levels elevated more than 1.5 times the upper limit of normal (ULN) within 7 days prior to enrollment
26. The absolute neutrophil count (ANC) < 2,000 per mm^3 within 7 days prior to enrollment
27. Platelet count less than 100,000 per mm^3 within 7 days prior to enrollment
28. More than 50% CD8+/ CD28- T-cells in peripheral blood
29. A calculated panel reactive antibody (cPRA) ≥20%, as determined by each participating site's laboratory
30. Positive pregnancy test in women of child bearing potential, currently breastfeeding, or planning to become pregnant during the timeframe of the study or follow-up period
31. Participation in any other studies with investigational drugs or regimens in the preceding year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Vincenti, M.D., Principal Investigator — University of California San Francisco School of Medicine: Transplantation; Sindhu Chandran, M.D., Study Chair — University of California San Francisco School of Medicine: Transplantation
Locations (7):
- United States (7):
  - University of Alabama School of Medicine: Transplantation, Birmingham, Alabama
  - University of California San Francisco School of Medicine: Transplantation, San Francisco, California
  - University of Colorado (UC) Health Transplant Center - Anschutz, Aurora, Colorado
  - Northwestern Memorial Hospital: Transplantation, Chicago, Illinois
  - University of Nebraska Medical Center: Transplantation, Omaha, Nebraska
  - Duke University Medical Center: Transplantation, Durham, North Carolina
  - Cleveland Clinic Foundation: Transplantation, Cleveland, Ohio

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation — https://www.niaid.nih.gov/about/dait
- See also: Clinical Trials in Organ Transplantation (CTOT) — http://www.ctotstudies.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 adult, kidney transplant candidates were enrolled across 4 US sites between December 2019 and March 2022. Of the 15 enrolled transplant candidates, 8 participants initiated treatment. The 7 participants who did not initiate study treatment were terminated because they did not meet eligibility criteria. Additionally, 9 donors were consented and enrolled across 3 US sites between December 2019 and August 2021.
Pre-assignment Details: Potential participants signed informed consent and enrolled before undergoing any study procedures. Screening criteria were evaluated to determine study eligibility. Participants were enrolled prior to transplantation. Living donors were asked to consent (at which point they were considered enrolled) for a single blood draw and minimal medical information.
Groups:
- Transplanted, Received Lulizumab: The participants underwent a transplant procedure and received rabbit anti-thymocyte globulin (rATG, Thymoglobulin) and methylprednisone and were initially maintained on tocilizumab and prednisone. Lulizumab pegol (BMS-931699) was administered on the day after transplantation and weekly until 3 months; after which it was replaced with belatacept every 4 weeks. MMF was started on the day after transplant. Everolimus was added 14 days post-transplant. MMF was discontinued once everolimus level was within therapeutic range. Tocilizumab was discontinued at 6 months post-transplant. Participants were then maintained on belatacept, everolimus, and prednisone.
- Screen Failure: Participants who failed screening.
- Enrolled Living Donor: Living donors of the prospective transplant recipient were consented and enrolled into the study.
Period: Overall Study
Arm/Group | Transplanted, Received Lulizumab | Screen Failure | Enrolled Living Donor
Started | 8 | 7 | 9
Completed | 6 | 0 | 9
Not Completed | 2 | 7 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Did Not Meet Eligibility Criteria | 0 | 7 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population, which includes the same subjects as the safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Transplanted, Received Lulizumab | Enrolled Living Donor | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.32) | 42.7 (10.26) | 46.2 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Who Remain Free of Biopsy-proven Acute T-cell Mediated or Antibody-mediated Rejection (as Defined by Banff Criteria) at 6 Months Post-transplantation.
Description: Acute T-cell mediated rejection was defined using the Banff 2007 criteria. Participants with a Banff grade of greater than or equal to 1A were determined to have met the endpoint. Severity is graded as 1A, 1B, 2A, 2B, or 3, with 1A being the mildest form of cellular rejection and 3 being the most severe form of cellular rejection. Antibody mediated rejection was defined as diffusely positive staining for C4d, presence of circulating anti-donor antibodies, and morphologic evidence of acute tissue injury. Clinical rejection occurring prior to 6 months, defined as treated rejection without biopsy confirmation was included as acute rejection with respect to the endpoint.
Time Frame: 6 months post-transplantation
Population: Intent-to-treat population, which includes the same subjects as the safety population, subset to participants who remained in the study in the 6 months following transplantation.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Transplanted, Received Lulizumab
Number analyzed (Participants) | 6
Proportion of participants | 0.500 [0.118 to 0.882]

2. Secondary Outcome: The Proportion of Participants Who Remain Free of Biopsy-proven Acute T-cell Mediated or Antibody-mediated Rejection (as Defined by Banff Criteria) at 12 Months Post-transplantation.
Description: Acute T-cell mediated rejection was defined using the Banff 2007 criteria. Participants with a Banff grade of greater than or equal to 1A were determined to have met the endpoint. Severity is graded as 1A, 1B, 2A, 2B, or 3, with 1A being the mildest form of cellular rejection and 3 being the most severe form of cellular rejection. Antibody mediated rejection was defined as diffusely positive staining for C4d, presence of circulating anti-donor antibodies, and morphologic evidence of acute tissue injury. Clinical rejection occurring prior to 12 months, defined as treated rejection without biopsy confirmation were included as acute rejection with respect to the endpoint.
Time Frame: 12 months post-transplantation
Population: Intent-to-treat population, which includes the same subjects as the safety population, subset to participants who remained in the study in the 12 months following transplantation.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Transplanted, Received Lulizumab
Number analyzed (Participants) | 6
Proportion of participants | 0.500 [0.118 to 0.882]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of first study mandated procedure until a subject completed study participation (either 24 months post-transplant or 12 months post-transplant, if entered into reduced follow-up) or until 30 days after they prematurely withdrew (without withdrawing consent) or was withdrawn from the study.
Groups:
- 'Transplanted/Received Lulizumab': 'The participants underwent a transplant procedure and received rabbit anti-thymocyte globulin (rATG, Thymoglobulin) and methylprednisone and were initially maintained on tocilizumab and prednisone. Lulizumab pegol (BMS-931699) was administered on the day after transplantation and weekly until 3 months; after which it was replaced with belatacept every 4 weeks. MMF was started on the day after transplant. Everolimus was added 14 days post-transplant. MMF was discontinued once everolimus level was within therapeutic range. Tocilizumab was discontinued at 6 months post-transplant. Participants were then maintained on belatacept, everolimus, and prednisone.'
- 'Enrolled Living Donor': 'Living donors of the prospective transplant recipient were consented and enrolled into the study.'
Arm/Group | 'Transplanted/Received Lulizumab' | 'Enrolled Living Donor'
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 8/8 | 0/9
Other Adverse Events (participants affected / at risk) | 5/8 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 'Transplanted/Received Lulizumab' (N=8) | 'Enrolled Living Donor' (N=9)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 3 (3) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (2) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (5) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Subcapsular renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 'Transplanted/Received Lulizumab' (N=8) | 'Enrolled Living Donor' (N=9)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella test positive (Investigations) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT04066114/Prot_SAP_002.pdf
  • Informed Consent Form: Donor ICF (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT04066114/ICF_000.pdf
  • Informed Consent Form: Recipient ICF (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT04066114/ICF_001.pdf